CLINICAL TRIAL: NCT01491165
Title: Safety and Efficacy of Umbilical Cord Mesenchyma Stem Cell Transplantation in Liver Cirrhosis Patients
Brief Title: Safety and Efficacy of Stem Cell Transplantation for Treatment of Liver Cirrhosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Collaborators: Xinjiang Armed Police Corps Hospital (Unknown); Taian Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-12-07 liver cirrhosis
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Other Surgical Procedures
Keywords: umbilical cord mesenchyma stem cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell transplantation therapy (Experimental): umbilical cord mesenchyma stem cell transplantation through interventional procedures do in liver cirrhosis patients.
  Interventions: Procedure: stem cell transplantation through interventional procedures

INTERVENTIONS:
Procedure: stem cell transplantation through interventional procedures — one time interventional procedures
  Other Names: umbilical cord mesenchyma stem cell transplantation

SUMMARY:
Mainstream of current treatment of liver cirrhosis is liver transplantation, but there are high cost, risk and immune rejection and other issues. Umbilical cord mesenchyma stem cell with self-and directed differentiation capacity can effectively rescue experimental liver failure and contribute to liver regeneration, which suggests the feasibility of stem cell transplantation therapy. In this study, the safety and efficacy of umbilical cord mesenchyma stem cell transplantation through interventional procedures in patients liver cirrhosis will be evaluated.

DETAILED DESCRIPTION:
This study included three research centers, each center were carried out 25 cases of liver cirrhosis in patients with stem cell transplantation. All the selection and exclusion criteria are same, data summary and analysis will be complete by the epidemiological commissioner.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of liver cirrhosis;
* Without hepatic encephalopathy;
* No ascites or have easily dissipated ascites;
* Value of bilirubin is less than 100;
* Value of albumin is greater than 16 g / L;
* Prothrombin time is less than 21 seconds;

Exclusion Criteria:

* Severe cardiovascular disease, and immunocompromised patients;
* Patients with localized lesions affecting graft infection;
* Coagulation disorders;
* Liver nodules more than 2cm or Liver cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
liver volume calculated by MRI | 3 days before transplantation, 6 and 12 months after transplantation
  Instrument:universal 1.5 Tesla superconducting MRI instrument. Slice thickness :2mm.

SECONDARY OUTCOMES:
liver biopsy | whinin 7 days before transplantation, 6 and 12 months after transplantation
  The result of liver biopsy judged by the expert.
gastroscopy | whinin 7 days before transplantation, 6 and 12 months after transplantation
  Observe and photograph the related varicose veins.
blood biochemistry | whinin 7 days before transplantation, 1,3,6 and 12 months after transplantation
  1. alanine aminotransferase
  2. aspartate aminotransferase
  3. gamma-glutamyltransferase(GGT)
  4. alkaline phosphatase
  5. total bilirubin
  6. direct bilirubin
  7. The total bile acid (TBA)
  8. serum cholinesterase (CHE)
  9. total cholesterol (TC)
  10. albumin
  11. the proportion of white balls
blood test | whinin 7 days before transplantation, 1,3,6 and 12 months after transplantation
  1. platelet count (PLT)
  2. mean platelet volume (MPV)
  3. platelet distribution width (PDW)
  4. platelet hematocrit (PCT)
  5. alpha feto protein(AFP)
liver enzyme fiber spectrum | whinin 7 days before transplantation, 1,3,6 and 12 months after transplantation
  1. laminin (LN)
  2. Ⅳ collagen detection (CIV)
  3. hyaluronic acid (HA)
  4. procollagen Ⅲ(PC Ⅲ)
coagulation | whinin 7 days before transplantation, 1,3,6 and 12 months after transplantation
  1. prothrombin time (PT)
  2. activated partial thromboplastin time (APTT)
  3. fibrinogen (FIB)
  4. thrombin time (TT)
portal vein and splenic vein measure | whinin 7 days before transplantation, 1,3,6 and 12 months after transplantation
  1. Portal vein diameter (Dpv);
  2. Portal vein maximum velocity (Vmaxpv);
  3. Portal vein blood flow per minute (Qpv);
  4. The splenic vein diameter (Dsv);
  5. Splenic vein maximum flow velocity (Vmaxsv);
  6. Splenic vein blood flow per minute (Qsv).

CONTACTS AND LOCATIONS:
Overall Officials: Yihua An, Study Director — Department of Stem Cell Transplantation, the General Hospital of Chinese People's Armed Police Force
Locations (1):
- Yihua An, Beijing, China